CLINICAL TRIAL: NCT04952259
Title: Evaluation of the Effect of Shexiang Tongxin Dripping Pills on Coronary Microcirculation in Patients With Acute Anterior Myocardial Infarction by Microcirculation Resistance Index
Brief Title: Effect of Shexiang Tongxin Dropping Pills on Microcirculation in Patients With AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2019480
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Pharmaceutical Preparations; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Shexiang Tongxin dripping pills + routine treatment
  Interventions: Drug: Shexiang Tongxin Dropping Pills + routine treatment
- Control group (Active Comparator): routine treatment
  Interventions: Procedure: routine treatment

INTERVENTIONS:
Drug: Shexiang Tongxin Dropping Pills + routine treatment — oral+percutaneous coronary intervention
  Other Names: drugs and surgery
  Arms: Intervention group
Procedure: routine treatment — percutaneous coronary intervention
  Other Names: surgery
  Arms: Control group

SUMMARY:
This study is a randomized, controlled clinical trial. Evaluation of microcirculation resistance by index of microcirculation resistance to explore the protective effect of Shexiang Tongxin dripping pills on microcirculation in patients with acute anterior myocardial infarction.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the best way to improve the prognosis of patients with acute myocardial infarction (AMI), and ischemia-reperfusion injury (I/R) can damage the vascular endothelium through complex mechanisms, leading to microcirculation dysfunction and aggravation myocardial damage and affect the prognosis. Cell and animal experiments have proved that Shexiang Tongxin Dropping Pill has anti-inflammatory, anti-oxidant, reducing I/R damage, reducing infarct size, improving peripheral muscle microcirculation, and improving coronary slow blood flow, but it lacks directive evidences of improved coronary microcirculation in AMI patients. The microcirculation resistance index (IMR) is a parameter to evaluate the microcirculation state obtained by the pressure/temperature guidewire during PCI, which can accurately and quantitatively reflect the patient's coronary microcirculation state. In this study, patients with acute anterior wall elevation ST-segment myocardial infarction (STEMI) who were prospectively selected for direct PCI treatment were randomly divided into treatment group and control group. The treatment group was given Shexiang Tongxin Dropping Pills before PCI and received direct PCI treatment, the control group only received direct PCI treatment. The IMR of the two groups was detected immediately after PCI, and the differences in IMR values, myocardial injury markers and cardiac function parameters between the two groups were analyzed. It is hoped to prove that Shexiang Tongxin dripping pills have coronary microcirculation protection in acute anterior wall elevation ST-segment myocardial infarction with undergoing direct PCI treatment, and the effect is rapid, so as to provide a basis for optimizing AMI treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, no gender limit;
* Anterior wall STEMI within 12 hours of onset (diagnostic criteria: ischemic chest pain lasting ≥30min; ST-segment elevation or new left bundle branch block in two or more adjacent leads on the ECG; with or without Elevated myocardial markers), emergency PCI treatment is planned;
* Infarct-related coronary vascular anatomy is suitable for PCI treatment;
* Agree and cooperate to participate in this research, and sign an informed consent form

Exclusion Criteria:

* Past history of myocardial infarction history;
* The arteries related to infarction have received PCI in the past;
* Past CABG history;
* Killip grade of cardiac function ≥ grade III or cardiogenic shock;
* Systolic blood pressure ≤90mmHg;
* Bradycardia, heart rate <60 beats/min, or atrioventricular block of degree II or more;
* Allergic to Shexiang Tongxin Dropping Pills
* Past history of asthma or severe COPD;
* Severe liver and kidney dysfunction;
* Participate in other clinical trials within 3 months;
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
IMR | detected immediately after percutaneous coronary intervention
  microcirculation resistance index

SECONDARY OUTCOMES:
Myocardial injury markers | 72 hours
  cardiac enzymes and troponin T

CONTACTS AND LOCATIONS:
Overall Officials: Liyun He, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No